CLINICAL TRIAL: NCT00505323
Title: Motor and Premotor Cortex Stimulation for Treatment of Secondary Focal Dystonia With Striato Pallidal Lesion : Evaluation of Safety and Effectiveness
Brief Title: Motor and Premotor Cortex Stimulation for Treatment of Secondary Focal Dystonia With Striato Palliadal Lesion : Evaluation of Safety and Effectiveness
Acronym: CORDYS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-A00100-53; PHRC N 2007 DURIF
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Focal Dystonia
Keywords: Cortex stimulation; Focal secondary Dystonia; Effectiveness; Quality of life improvement; Focal dystonias secondary to central grey nuclei lesions
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Device: Implantation of neurostimulators and their auxiliary components — Implantation neurostimulators and their auxiliary components :
  Stimulateur KINETRA TM modèle 7428, Electrode Resume II modèle 3587A, Extension kit DBS 7482

SUMMARY:
Dystonia is a neurological movement disorder in which sustained muscle contractions cause twisting and repetitive movements or abnormal postures. This disease is very heterogeneous and can have many causes. Current treatments (drugs, pallidal stimulation) improve primary generalized dystonias; however they are ineffective for focal dystonias following brain damage.

Cortex stimulation is a present and effective technique used in the treatment of chronic pain and could represent an interesting strategy to treat focal dystonias. This is the aim of the present study.

DETAILED DESCRIPTION:
Pilot study included 6 centres (Clermont-Ferrand, Bordeaux, Paris, Créteil, Lyon and Grenoble)

Study progress :

* 3 months to 1 month before chirurgical intervention : selection of patient that could be included in the protocol.
* 15 days to 8 days before chirurgical intervention : inclusion visit.
* Operating phase : under anaesthesia, implantation of the neurostimulator and its components, and adjustment of stimulation parameters.
* 1 month after chirurgical intervention : checking that all is fine (detection of undesirable events)
* 2 months to 5 months after chirurgical intervention: randomization (double blind): the stimulator is put on position On or OFF
* 5 months after chirurgical intervention : Stimulators of all patients are stopped for one month whatever the group they belong.
* 6 months to 9 months after chirurgical intervention: Stimulatiors are put on position On or OFF (cross over with the first period).
* 9 months to 13 months after chirurgical intervention: Stimulators of all patients are started for four months whatever the group they belong.
* 13 months after chirurgical intervention : study end

ELIGIBILITY:
Inclusion Criteria:

* Age : >18 years and < 65 years
* Evolution time of dystonia > 1 year
* Clinical stability of dystonia = 1 year
* Secondary dystonia due to a focal lesion (vascular or anoxic) of central grey nuclei
* Inefficiency of others treatments (anticholinergic, benzodiazepine, neuroleptique, botulinum toxin, etc.)
* Stability of treatment >3 months
* Agreement of patients
* Affiliation to social security

Exclusion Criteria:

* Significant heart vascular disease; significant respiratory, metabolic, renal or hepatic diseases
* Significant clinical and biological anomalies
* Disease or treatment in favour in bleeding
* Sever cognitive disorders
* Psychiatric evolutionary pathology
* Counter-indication during inclusion examination
* Chirurgical counter-indication
* Pregnant women ou women who nurse
* Person who participate to an other study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of dystonia by using the validated "Burke Fahn and Marsden (1985)" dystonia rating scale | before the chirurgical intervention and 2, 5, 6, 9 and 13 months after

SECONDARY OUTCOMES:
Evaluation of spasticity (Ashworth), of akinesy (Tapping score), of pain (EVA test), of quality of life (SF 36 scale) and of undesirable events. | before the chirurgical intervention and 2, 5, 6, 9 and 13 months after

CONTACTS AND LOCATIONS:
Overall Officials: Franck DURIF, Pr, Principal Investigator